CLINICAL TRIAL: NCT05144074
Title: CD62P(P-selectin) as a Marker of Assessment of Platelet Storage Lesion(PSL)in Platelet Concentrates
Brief Title: Assessment of Platelet Storage Lesion(PSL)in Platelet Concentrates
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Merna Mamdoh Ayad Benyamen, resident, Assiut University
Other Study IDs: platelet storage lesion
Record Dates: First submitted 2021-11-21; First posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Platelet Storage Lesion(PSL)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-filtered platelet concentrates (NF-PC group).: In NF-PC group, 90 whole blood units were collected with Tripple blood bags, Six NF-PCs were pooled together and stored in a horizonal shaker at 20 ± 2C for 5 days .
- leukocyte-depleted platelet concentrates (LD-PC group).: In LD-PC group, another 90 whole blood units were collected using Whole Blood Filter Saving Platelets (WB-SP) bags with an integrated leukoreduction filter

SUMMARY:
The aim of this study to assess platelet activation during 5 days storage of platelet concentrates prepared by different techinques .

DETAILED DESCRIPTION:
Platelet transfusion is a lifesaving procedure that is carried out to prevent bleeding or stop ongoing bleeding in patients with low platelet count or functional platelet disorders. There are minimum thresholds at which platelets are transfused in these patients, as not all low levels of platelet warrants a transfusion. Platelet is a scarce resource as processing, preparing, and transfusing it requires a great deal of precision and effort to maintain a certain quality. This activity highlights the use of platelet transfusion by the interprofessional team (1).

Platelets play an integral role in hemostasis by its response to vascular injury. The relevance of platelet component therapy was better understood in the 1950s and 1960s when severe and fatal hemorrhagic complications of chemotherapy in leukemia were studied

The collected blood units were randomly assigned to two groups:

1. Non-filtered platelet concentrates (NF-PC group).
2. leukocyte-depleted platelet concentrates (LD-PC group). P-selectin (CD62p) is a type of glycoprotein stored in the Weibel-Palade bodies of vascular endothelial cells and platelet α-granules. Activated CD62P is a transmembrane protein expressed on the platelet surface. During platelet activation, the expression of CD62P on the surface of the cell membrane is dramatically increased in PCs without leukocyte depletion, due to the presence of WBCs and cytokines ,and is accompanied by an increase in the expression level of plasma soluble CD62

ELIGIBILITY:
Inclusion Criteria:

* Donors who met criteria of Egyptian National Transfusion services
* Donors who had not taken any antiplatelet drugs for two weeks prior to donation
* pre-collection platelet count ≥200×109 /L.
* Blood grouping.
* Serological assays for all blood donors (HBsAgs, HCV antibodies, HIV Ag/Ab Syphilis antibodies) on Architect i 2000 SR or Centaur XPT (chemoluminescence).

Exclusion Criteria:

* Donors who not met criteria of Egyptian National Transfusion services
* Donors who had taken any antiplatelet drugs for two weeks prior to donation
* pre-collection platelet count <200×109 /L.
* Reactive serology

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: All gender fullfilling inclusion criteria are participating in this study ,
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
assess platelet activation . | baseline
  assess platelet activation during 5 days storage of platelet concentrates prepared by different techinques .

SECONDARY OUTCOMES:
CD62p assessment . | baseline
  CD62p assessment of platelet storage lesion(PSL)in platelet concentrates .

REFERENCES:
- [Background] Freireich EJ. Origins of platelet transfusion therapy. Transfus Med Rev. 2011 Jul;25(3):252-6. doi: 10.1016/j.tmrv.2011.01.003. Epub 2011 Mar 2. PMID 21371858
- [Background] Kaushansky K. The molecular mechanisms that control thrombopoiesis. J Clin Invest. 2005 Dec;115(12):3339-47. doi: 10.1172/JCI26674. PMID 16322778
- [Background] Solves Alcaina P. Platelet Transfusion: And Update on Challenges and Outcomes. J Blood Med. 2020 Jan 24;11:19-26. doi: 10.2147/JBM.S234374. eCollection 2020. PMID 32158298
- [Background] Cines DB, Levine LD. Thrombocytopenia in pregnancy. Hematology Am Soc Hematol Educ Program. 2017 Dec 8;2017(1):144-151. doi: 10.1182/asheducation-2017.1.144. PMID 29222249